CLINICAL TRIAL: NCT06080594
Title: Exercise-mediated Rescue of Mitochondrial Derangements Driving Insulin Resistance in Humans (EX-MITO-DYS-IR)
Brief Title: Exercise-mediated Rescue of Mitochondrial Dysfunctions Driving Insulin Resistance
Acronym: EX-MITO-DYS-IR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Matteo Fiorenza, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EX-MITO-DYS-IR
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Mitochondrial Myopathies; Mitochondrial Diseases; Mitochondrial Disorders
Keywords: Mitochondrial disease; Muscle metabolism; Insulin resistance; Exercise training; Mitochondrial dysfunction
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: In a within-subject parallel-group longitudinal design, participants sustain an exercise training intervention with one leg, while the contralateral leg serves as an inactive control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise leg (Experimental): High-intensity exercise training for one leg
  Interventions: Behavioral: High-intensity exercise training
- Control leg (No Intervention): No exercise training for the controlateral leg

INTERVENTIONS:
Behavioral: High-intensity exercise training — Eight sessions of high-intensity interval exercise using a single-leg cycle ergometer are conducted on separate days over a 2-week period.
  Other Names: High-intensity interval training
  Arms: Exercise leg

SUMMARY:
The overarching aim of this intervention study is to interrogate the interconnection between the muscle mitochondrial adaptations and the changes in muscle insulin sensitivity elicited by exercise training in individuals harbouring pathogenic mitochondrial DNA mutations associated with an insulin-resistant phenotype.

In a within-subject parallel-group longitudinal design, participants will undergo an exercise training intervention with one leg, while the contralateral leg will serve as an inactive control. After the exercise intervention, patients will attend an experimental trial including:

* A hyperinsulinemic-euglycemic clamp combined with measurements of femoral artery blood flow and arteriovenous difference of glucose
* Muscle biopsy samples

DETAILED DESCRIPTION:
Background: Peripheral insulin resistance is a major risk factor for metabolic diseases such as type 2 diabetes. Skeletal muscle accounts for the majority of insulin-stimulated glucose disposal, hence restoring insulin action in skeletal muscle is key in the prevention of type 2 diabetes. Mitochondrial dysfunction is implicated in the etiology of muscle insulin resistance. Also, as mitochondrial function is determined by its proteome quantity and quality, alterations in the muscle mitochondrial proteome may play a critical role in the pathophysiology of insulin resistance. However, insulin resistance is multifactorial in nature and whether mitochondrial derangements are a cause or a consequence of impaired insulin action is unclear. In recent years, the study of humans with genetic mutations has shown enormous potential to establish the mechanistic link between two physiological variables; indeed, if the mutation has a functional impact on one of those variables, then the direction of causality can be readily ascribed. Mitochondrial myopathies are genetic disorders of the mitochondrial respiratory chain affecting predominantly skeletal muscle. Mitochondrial myopathies are caused by pathogenic mutations in either nuclear or mitochondrial DNA (mtDNA), which ultimately lead to mitochondrial dysfunction. Although the prevalence of mtDNA mutations is just 1 in 5,000, the study of patients with mtDNA defects has the potential to provide unique information on the pathogenic role of mitochondrial derangements that is disproportionate to the rarity of affected individuals. The m.3243A>G mutation in the MT-TL1 gene encoding the mitochondrial leucyl-tRNA 1 gene is the most common mutation leading to mitochondrial myopathy in humans. The m.3243A>G mutation is associated with impaired glucose tolerance and insulin resistance in skeletal muscle. Most importantly, insulin resistance precedes impairments of β-cell function in carriers of the m.3243A>G mutation, making these patients an ideal human model to study the causative nexus between muscle mitochondrial dysfunction and insulin resistance. Exercise training is a potent stimulus to enhance muscle insulin action, improve mitochondrial function, and promote mitochondrial proteome remodeling. Accordingly, rescue of mitochondrial dysfunction has been proposed to play a role in the insulin-sensitizing effect of exercise. Yet, numerous mechanisms may contribute to the pathophysiology of insulin resistance and the beneficial effects of exercise may be linked to amelioration of multiple factors, thus challenging the interpretation of the functional significance of improved muscle mitochondrial function per se. Nevertheless, since mitochondrial dysfunction is likely the primary cause of muscle insulin resistance in carriers of the m.3243A>G mutation, prospective studies including an in-depth analysis of the mitochondrial adaptations elicited by exercise training in this cohort of patients may offer a unique opportunity to identify those mitochondrial derangements that, once rescued, drive enhancements in insulin sensitivity.

Objective: To study the effects of exercise training on muscle insulin sensitivity, muscle mitochondrial function, and the muscle mitochondrial proteome in individuals harboring pathogenic mitochondrial DNA (mtDNA) mutations associated with an insulin-resistant phenotype.

Study design: Within-subject parallel-group longitudinal study in individuals with pathogenic mtDNA mutations undergoing an exercise training intervention with one leg (contralateral leg as inactive control).

Endpoint: Differences between the trained and the untrained leg.

ELIGIBILITY:
Inclusion Criteria:

* Known m.3243A>G mutation in the MT-TL1 gene encoding the mitochondrial leucyl-tRNA 1 gene
* Other known mtDNA point mutations

Exclusion Criteria:

* Use of antiarrhythmic medications or other medications which, in the opinion of the investigators, have the potential to affect outcome measures.
* Diagnosed severe heart disease, dysregulated thyroid gland conditions, or other dysregulated endocrinopathies, or other conditions which, in the opinion of the investigators, have the potential to affect outcome measures.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | 90-150 minutes after initiation of a hyperinsulinemic euglycemic clamp
  Insulin-stimulated muscle glucose uptake is determined by the hyperinsulinemic-euglycemic clamp method integrated with measurements of femoral artery blood flow and arteriovenous difference of glucose
Muscle mitochondrial respiration | Baseline
  Mitochondrial O2 flux is measured by high-resolution respirometry in permeabilized fibers from muscle biopsy samples
Muscle mitochondrial reactive oxygen species (ROS) production | Baseline
  Mitochondrial H2O2 emission rates are measured by high-resolution fluorometry in permeabilized fibers from muscle biopsy samples
Muscle mitochondrial proteome | Baseline
  Mitochondrial proteome signatures are determined by mass spectrometry-based proteomics in muscle biopsy samples

SECONDARY OUTCOMES:
Muscle mtDNA heteroplasmy | Baseline
  mtDNA mutation load is measured in muscle biopsy samples from the patients with mitochondrial myopathy
Muscle insulin signaling | Before (baseline) and 150 minutes after initiation of the hyperinsulinemic-euglycemic clamp
  Insulin-mediated changes in the abundance of (phosphorylated) proteins modulating insulin action are measured by immunoblotting in muscle and fat biopsy samples
Muscle integrated stress response signaling proteins | Baseline
  Abundance of (phosphorylated) proteins governing the integrated stress response pathway is measured by immunoblotting in muscle biopsy samples.
Muscle integrated stress response genes | Baseline
  mRNA content of genes governing the integrated stress response pathway is measured by Real-Time PCR in muscle biopsy samples.
Muscle release of FGF21 and GDF15 | Before (baseline) and 0-150 minutes after initiation of the hyperinsulinemic-euglycemic clamp
  Skeletal muscle production of FGF21 and GDF15 is determined by measurements of femoral artery blood flow and arteriovenous difference of plasma FGF21 and GDF15
Whole-body insulin sensitivity | 90-150 minutes after initiation of a hyperinsulinemic euglycemic clamp
  Whole-body insulin sensitivity is determined by the hyperinsulinemic-euglycemic clamp method

OTHER OUTCOMES:
Leg muscle mass | Baseline
  Leg muscle mass is determined by dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Fiorenza, Ph.D., Principal Investigator — Rigshospitalet, Denmark; John Vissing, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFronzo RA, Ferrannini E. Insulin resistance. A multifaceted syndrome responsible for NIDDM, obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Diabetes Care. 1991 Mar;14(3):173-94. doi: 10.2337/diacare.14.3.173. PMID 2044434
- [Background] DeFronzo RA, Simonson D, Ferrannini E. Hepatic and peripheral insulin resistance: a common feature of type 2 (non-insulin-dependent) and type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1982 Oct;23(4):313-9. doi: 10.1007/BF00253736. PMID 6754515
- [Background] DeFronzo RA, Gunnarsson R, Bjorkman O, Olsson M, Wahren J. Effects of insulin on peripheral and splanchnic glucose metabolism in noninsulin-dependent (type II) diabetes mellitus. J Clin Invest. 1985 Jul;76(1):149-55. doi: 10.1172/JCI111938. PMID 3894418
- [Background] Diaz-Vegas A, Sanchez-Aguilera P, Krycer JR, Morales PE, Monsalves-Alvarez M, Cifuentes M, Rothermel BA, Lavandero S. Is Mitochondrial Dysfunction a Common Root of Noncommunicable Chronic Diseases? Endocr Rev. 2020 Jun 1;41(3):bnaa005. doi: 10.1210/endrev/bnaa005. PMID 32179913
- [Background] Hesselink MK, Schrauwen-Hinderling V, Schrauwen P. Skeletal muscle mitochondria as a target to prevent or treat type 2 diabetes mellitus. Nat Rev Endocrinol. 2016 Nov;12(11):633-645. doi: 10.1038/nrendo.2016.104. Epub 2016 Jul 22. PMID 27448057
- [Background] Parish R, Petersen KF. Mitochondrial dysfunction and type 2 diabetes. Curr Diab Rep. 2005 Jun;5(3):177-83. doi: 10.1007/s11892-005-0006-3. PMID 15929863
- [Background] Zabielski P, Lanza IR, Gopala S, Heppelmann CJ, Bergen HR 3rd, Dasari S, Nair KS. Altered Skeletal Muscle Mitochondrial Proteome As the Basis of Disruption of Mitochondrial Function in Diabetic Mice. Diabetes. 2016 Mar;65(3):561-73. doi: 10.2337/db15-0823. Epub 2015 Dec 30. PMID 26718503
- [Background] Petersen MC, Shulman GI. Mechanisms of Insulin Action and Insulin Resistance. Physiol Rev. 2018 Oct 1;98(4):2133-2223. doi: 10.1152/physrev.00063.2017. PMID 30067154
- [Background] O'Rahilly S. "Treasure Your Exceptions"-Studying Human Extreme Phenotypes to Illuminate Metabolic Health and Disease: The 2019 Banting Medal for Scientific Achievement Lecture. Diabetes. 2021 Jan;70(1):29-38. doi: 10.2337/dbi19-0037. PMID 33355307
- [Background] Saleheen D, Natarajan P, Armean IM, Zhao W, Rasheed A, Khetarpal SA, Won HH, Karczewski KJ, O'Donnell-Luria AH, Samocha KE, Weisburd B, Gupta N, Zaidi M, Samuel M, Imran A, Abbas S, Majeed F, Ishaq M, Akhtar S, Trindade K, Mucksavage M, Qamar N, Zaman KS, Yaqoob Z, Saghir T, Rizvi SNH, Memon A, Hayyat Mallick N, Ishaq M, Rasheed SZ, Memon FU, Mahmood K, Ahmed N, Do R, Krauss RM, MacArthur DG, Gabriel S, Lander ES, Daly MJ, Frossard P, Danesh J, Rader DJ, Kathiresan S. Human knockouts and phenotypic analysis in a cohort with a high rate of consanguinity. Nature. 2017 Apr 12;544(7649):235-239. doi: 10.1038/nature22034. PMID 28406212
- [Background] DiMauro S. Mitochondrial myopathies. Curr Opin Rheumatol. 2006 Nov;18(6):636-41. doi: 10.1097/01.bor.0000245729.17759.f2. PMID 17053512
- [Background] Gorman GS, Schaefer AM, Ng Y, Gomez N, Blakely EL, Alston CL, Feeney C, Horvath R, Yu-Wai-Man P, Chinnery PF, Taylor RW, Turnbull DM, McFarland R. Prevalence of nuclear and mitochondrial DNA mutations related to adult mitochondrial disease. Ann Neurol. 2015 May;77(5):753-9. doi: 10.1002/ana.24362. Epub 2015 Mar 28. PMID 25652200
- [Background] Elliott HR, Samuels DC, Eden JA, Relton CL, Chinnery PF. Pathogenic mitochondrial DNA mutations are common in the general population. Am J Hum Genet. 2008 Aug;83(2):254-60. doi: 10.1016/j.ajhg.2008.07.004. PMID 18674747
- [Background] Frederiksen AL, Jeppesen TD, Vissing J, Schwartz M, Kyvik KO, Schmitz O, Poulsen PL, Andersen PH. High prevalence of impaired glucose homeostasis and myopathy in asymptomatic and oligosymptomatic 3243A>G mitochondrial DNA mutation-positive subjects. J Clin Endocrinol Metab. 2009 Aug;94(8):2872-9. doi: 10.1210/jc.2009-0235. Epub 2009 May 26. PMID 19470628
- [Background] Lindroos MM, Majamaa K, Tura A, Mari A, Kalliokoski KK, Taittonen MT, Iozzo P, Nuutila P. m.3243A>G mutation in mitochondrial DNA leads to decreased insulin sensitivity in skeletal muscle and to progressive beta-cell dysfunction. Diabetes. 2009 Mar;58(3):543-9. doi: 10.2337/db08-0981. Epub 2008 Dec 10. PMID 19073775
- [Background] Deshmukh AS, Steenberg DE, Hostrup M, Birk JB, Larsen JK, Santos A, Kjobsted R, Hingst JR, Scheele CC, Murgia M, Kiens B, Richter EA, Mann M, Wojtaszewski JFP. Deep muscle-proteomic analysis of freeze-dried human muscle biopsies reveals fiber type-specific adaptations to exercise training. Nat Commun. 2021 Jan 12;12(1):304. doi: 10.1038/s41467-020-20556-8. PMID 33436631
- [Background] Meex RC, Schrauwen-Hinderling VB, Moonen-Kornips E, Schaart G, Mensink M, Phielix E, van de Weijer T, Sels JP, Schrauwen P, Hesselink MK. Restoration of muscle mitochondrial function and metabolic flexibility in type 2 diabetes by exercise training is paralleled by increased myocellular fat storage and improved insulin sensitivity. Diabetes. 2010 Mar;59(3):572-9. doi: 10.2337/db09-1322. Epub 2009 Dec 22. PMID 20028948